CLINICAL TRIAL: NCT03205618
Title: Effectiveness of Daclatasvir-Containing Regimens in Patients Treated in Real-Life Setting in Kingdom of Saudi Arabia (KSA), United Arab Emirates (UAE) and Qatar
Brief Title: A Retrospective, Observational Study on the Effectiveness of Daclatasvir-Containing Regimens in Patients in KSA, UAE and Qatar
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: AI444-382
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- daclatasvir patients in KSA, UAE, and Qatar: patients treated with daclatasvir-containing regimens in KSA, UAE, and Qatar
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
The study will provide safety and efficacy information among patients receiving daclatasvir. It will describe daclatasvir prescribing patterns and provide a clinical profile of patients receiving the treatment in KSA, UAE, and Qatar.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients greater than or equal to 18 years of age
* Diagnosed with chronic hepatitis C
* Ended treatment with daclatasvir-containing regimen no later than 01-Oct-2015

Exclusion Criteria:

* Use of a daclatasvir-containing regimen in a clinical trial setting

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll all patients initiating a new daclatasvir-containing HCV treatment, regardless of treatment history and previous treatment response from availability of the drug on country markets up to 01-Oct-2015.
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2016-04-26 (Actual); Primary Completion 2017-06-27 (Actual); Study Completion 2017-06-27 (Actual)

PRIMARY OUTCOMES:
Number of participants achieving sustained virological response 12 weeks post-treatment (SVR12) | 12 weeks after the last dose of study treatment
  Patients will be considered to have achieved SVR12 if they have a documented undetectable viral load on or after Week 12 following the end of treatment.

SECONDARY OUTCOMES:
Distribution of SVR12 by Treatment Regimen | 12 weeks after the last dose of study treatment
  Defined as any daclatasvir containing regimen. Subgroups include: daclatasvir + sofosbuvir; daclatasvir + sofosbuvir + RBV; daclatasvir + simeprevir; daclatasvir + simeprevir + ribavirin.
Distribution of SVR12 by Country | 12 weeks after the last dose of study treatment
  Defined as the country where treatment with a daclatasvir containing regimen was initiated. Subgroups include Saudi Arabia, UAE, and Qatar.
Distribution of SVR12 by Genotype | 12 weeks after the last dose of study treatment
  Subgroups genotype 3 and genotype 4
Distribution of SVR12 by HCV-Treatment Experience | 12 weeks after the last dose of study treatment
  Subgroups include patients in which prior treatment with IFN and RBV has failed; prior treatment with IFN, RBV and telaprevir or boceprevir has failed; previous treatment with IFN, RBV and simeprevir has failed; previous treatment with sofosbuvir and RBV has failed.
Distribution of SVR12 by HIV co-infection | 12 weeks after the last dose of study treatment
  Subgroup defined as HIV diagnosis prior to the initiation of daclatasvir containing regimen.
Distribution of SVR12 by previous liver transplantation | 12 weeks after the last dose of study treatment
  Subgroup defined by patients undergoing a liver transplant for any cause prior to the initiation of a daclatasvir containing regimen
Incidence of Serious Adverse Events (SAE) | Up to 12 months
  Measured by number of patients reporting SAEs
Incidence of Adverse Events leading to discontinuation | Up to 12 months
  Measured by number of patients reporting AEs that result in treatment discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- Saudi Arabia (3):
  - Local Institution, Doha
  - Local Institution, Jeddah
  - Local Institution, Riyadh-11211

REFERENCES:
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx